CLINICAL TRIAL: NCT00675792
Title: A Multi-center, Randomized, Parallel Group, Comparative, Active Controlled, Safety-assessor Blinded, Anesthesiologist-TOF-Watch® SX Blinded Trial Comparing T4/T1 Ratio at Time of Tracheal Extubation Using 4 mg/kg Sugammadex Administered at 1-2 PTCs or Better After the Last Dose of Rocuronium Bromide to 50 µg/kg Neostigmine Administered as Per Standard of Care in Adult Subjects Undergoing Elective Open Abdominal Procedures Requiring Neuromuscular Blockade Reversal
Brief Title: Comparison of Sugammadex Administered at 1-2 Post Tetanic Counts (PTCs) or Better With Neostigmine Administered as Per Standard of Care to Reverse Rocuronium-Induced Neuromuscular Blockade in Adults Undergoing Elective Open Abdominal Procedure (19.4.334) (P05774)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P05774; 19.4.334 (Other: Merck)
Record Dates: First submitted 2008-05-07; First posted 2008-05-12 (Estimated); Results first posted 2013-07-11 (Estimated); Last update posted 2015-03-13 (Estimated); Status verified 2015-02

CONDITIONS: Anesthesia
MeSH Terms: interventions — Sugammadex; Neostigmine; Rocuronium

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sugammadex (Experimental): 4 mg/kg sugammadex
  Interventions: Drug: Sugammadex; Drug: Rocuronium
- Neostigmine (Active Comparator): 50 µg/kg neostigmine
  Interventions: Drug: Neostigmine; Drug: Rocuronium

INTERVENTIONS:
Drug: Sugammadex — Participants received 4 mg/kg sugammadex at 1-2 Post Tetanic Counts (PTCs) or better after the last dose of rocuronium bromide.
  Other Names: Org 25969; SCH 900616; MK-8616; Bridion®
  Arms: Sugammadex
Drug: Neostigmine — Participants received 50 µg/kg neostigmine combined with 10 µg/kg glycopyrrolate after the last dose of rocuronium bromide as per standard of care.
  Other Names: Prostigmin®
  Arms: Neostigmine
Drug: Rocuronium — Participants received a single intubation bolus dose of 0.6 mg/kg rocuronium bromide, followed if necessary to maintain neuromuscular blockade by one or more single bolus dose(s) of 0.15 mg/kg rocuronium bromide.
  Other Names: Rocuronium bromide; Esmeron®

SUMMARY:
The primary purpose of this study is to compare the incidence of

residual neuromuscular blockade at the time of tracheal extubation after reversal of rocuronium bromide-induced neuromuscular blockade by 4 mg/kg sugammadex with that of 50 µg/kg neostigmine. Residual neuromuscular blockade is defined as the fourth twitch to first twitch (T4/T1) ratio of

< 0.90.

DETAILED DESCRIPTION:
Undetected residual neuromuscular blockade is common in the post-anesthesia care

unit (PACU). In fact, 16%-42% of patients receiving intermediate-acting muscle

relaxants in the operating room have T4/T1 ratios <0.7-0.8 in the PACU. Respiratory and pharyngeal muscle function can be adversely affected during minimal neuromuscular blockade. Studies in awake volunteers and surgical patients have demonstrated that T4/T1 ratios of 0.7 - 0.9 are associated with impaired airway protective reflexes, upper airway obstruction, a decreased hypoxic ventilatory response, and post-operative hypoxemia. The incidence and severity of residual neuromuscular blockade at the time of tracheal extubation will be evaluated to determine how these influence the length of stay in the operating room and PACU.

ELIGIBILITY:
Inclusion Criteria:

* male or females who are >= 18 and <= 65 years of age
* classified by the American Society of Anesthesiologists (ASA) as Class 1 or 2 or 3;
* Body Mass Index (BMI) of <35 kg/m^2;
* is scheduled to undergo an elective open abdominal surgical procedure under general anesthesia requiring neuromuscular relaxation using rocuronium bromide (maintenance of neuromuscular blockade if required) for endotracheal intubation and requiring neuromuscular blockade reversal;
* is scheduled to undergo a surgical procedure in a position that does not interfere with the use of TOF-Watch® SX;
* is scheduled to undergo an elective open abdominal procedure expected to last <=4 hours (from start of skin incision to end of last stitch of the skin);
* have given written informed consent.

Exclusion Criteria:

* participants for whom a difficult intubation is expected because of anatomical malformations;
* is known or suspected to have neuromuscular disorders that may impair neuromuscular blockade;
* is known or suspected to have significant renal dysfunction (e.g., creatinine clearance < 30 mL/min) ;
* is known or suspected to have significant hepatic dysfunction;
* is known or suspected to have a (family) history of malignant hyperthermia;
* is known or suspected to have an allergy to opioids, muscle relaxants or other medications used during general anesthesia;
* participants for whom the use of neostigmine and/or glycopyrrolate may be contraindicated;
* participants for whom a pre-established need for postoperative intensive care admission is expected;
* pregnant or breast-feeding females;
* have participated in a previous sugammadex clinical trial;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-05; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

REFERENCES:
- [Result] Sabo D, Jones RK, Berry J, Sloan T, Chen J-Y, Morte JB, Groudine S. Residual neuromuscular blockade at extubation: a randomized comparison of sugammadex and neostigmine reversal of rocuronium-induced blockade in patients undergoing abdominal surgery. J Anesthe Clin Res. 2011;2:140.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sugammadex | Neostigmine
Started | 51 | 49
Completed | 51 | 49
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sugammadex | Neostigmine | Total
Number analyzed (Participants) | 51 | 49 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (11) | 52 (9) | 51 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 31 | 60
  Male | 22 | 18 | 40

OUTCOME MEASURES:

1. Primary Outcome: Residual Neuromuscular Blockade Evidenced by T4/T1 Ratio at the Time of Tracheal Extubation
Description: Neuromuscular function was monitored by applying repetitive Train-Of-Four (TOF) electrical stimulations to the ulnar nerve every 15 seconds, and assessing twitch response at the adductor pollicis muscle with a TOF-Watch® SX. The magnitudes (heights) of the first and fourth twitches (T1 and T4) were used to calculate the T4/T1 ratio, where a higher T4/T1 ratio indicates a greater recovery from neuromuscular blockade, with a value of 1.0 indicating complete recovery. After anesthesia, when neuromuscular function was expected to be fully recovered, tracheal extubation was performed, at which time the T4/T1 ratio was measured, with any missing recovery times imputed.
Time Frame: Up to the first 24 hours after tracheal extubation
Population: Intent to treat (ITT) group consisting of all randomized participants who were treated with sugammadex or neostigmine and had at least one efficacy measurement. Three participants treated with neostigmine did not have at least one efficacy measurement, and hence were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: T4/T1 Ratio
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 51 | 46
T4/T1 Ratio | 1.02 (0.15) | 0.78 (0.24)

2. Secondary Outcome: Number of Participants With Post-operative Complications
Description: Post-operative complications include any of the following: procedural pain, nausea, vomiting, incision-site pain, constipation, headache, pyrexia, dizziness and pruritus.
Time Frame: Up to 7 days after surgery
Population: All subjects treated (AST) group consisting of randomized participants who were treated with sugammadex or neostigmine
Measure: Number; unit: participants
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 51 | 49
participants | 51 | 49

3. Secondary Outcome: Number of Participants With Evidence of Possible Interaction of Sugammadex With Endogenous Compounds or Exogenous Compounds Other Than Rocuronium Bromide
Description: Evidence of adverse events due to a possible interaction of sugammadex with exogenous compounds or endogenous compounds other than rocuronium was recorded.
Time Frame: Up to 7 days after surgery
Population: All subjects treated (AST) group consisting of randomized participants who were treated with sugammadex or neostigmine
Measure: Number; unit: participants
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 51 | 49
participants | 0 | 0

4. Secondary Outcome: Time From Start of Administration of Investigational Medicinal Product (IMP) to Recovery of the T4/T1 Ratio to 0.9
Description: Neuromuscular function was monitored by applying repetitive TOF electrical stimulations to the ulnar nerve every 15 seconds, and assessing T1 and T4 twitch response at the adductor pollicis muscle with a TOF-Watch® SX. Nerve stimulation was continued until the T4/T1 ratio, which indicates the extent of recovery from neuromuscular blockade, achieved a ratio of 0.9, with imputed data included.
Time Frame: Up to 1 hour after treatment
Population: ITT group consisting of all randomized participants who were treated with sugammadex or neostigmine and had at least one efficacy measurement. Three participants treated with neostigmine did not have at least one efficacy measurement, and hence were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 51 | 46
Minutes | 2.53 (1.18) | 7.95 (6.92)

5. Secondary Outcome: Time From Start of Administration of IMP to Recovery of the T4/T1 Ratio to 0.8
Description: Neuromuscular function was monitored by applying repetitive TOF electrical stimulations to the ulnar nerve every 15 seconds, and assessing T1 and T4 twitch response at the adductor pollicis muscle with a TOF-Watch® SX. Nerve stimulation was continued until the T4/T1 ratio, which indicates the extent of recovery from neuromuscular blockade, achieved a ratio of 0.8, with imputed data included.
Time Frame: Up to 1 hour after treatment
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 51 | 46
Minutes | 1.87 (0.82) | 6.18 (5.73)

6. Secondary Outcome: Time From Start of Administration of IMP to Recovery of the T4/T1 Ratio to 0.7
Description: Neuromuscular function was monitored by applying repetitive TOF electrical stimulations to the ulnar nerve every 15 seconds, and assessing T1 and T4 twitch response at the adductor pollicis muscle with a TOF-Watch® SX. Nerve stimulation was continued until the T4/T1 ratio, which indicates the extent of recovery from neuromuscular blockade, achieved a ratio of 0.7, with imputed data included.
Time Frame: Up to 1 hour after treatment
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 51 | 46
Minutes | 1.60 (0.72) | 4.98 (4.98)

ADVERSE EVENTS:
Time Frame: Up to 7 days after administration of IMP
Arm/Group | Sugammadex | Neostigmine
Serious Adverse Events (participants affected / at risk) | 4/51 | 6/49
Other Adverse Events (participants affected / at risk) | 51/51 | 49/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sugammadex (N=51) | Neostigmine (N=49)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 2 (2)
Pelvic abscess (Infections and infestations) | 0 (0) | 1 (1)
Wound infection staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Anastomotic leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sugammadex (N=51) | Neostigmine (N=49)
Abdominal distension (Gastrointestinal disorders) | 5 (5) | 1 (1)
Constipation (Gastrointestinal disorders) | 6 (6) | 6 (6)
Flatulence (Gastrointestinal disorders) | 4 (4) | 3 (3)
Ileus (Gastrointestinal disorders) | 0 (0) | 3 (3)
Nausea (Gastrointestinal disorders) | 26 (26) | 24 (24)
Vomiting (Gastrointestinal disorders) | 9 (9) | 11 (11)
Pyrexia (General disorders) | 7 (7) | 2 (2)
Incision site pain (Injury, poisoning and procedural complications) | 7 (7) | 9 (9)
Procedural hypertension (Injury, poisoning and procedural complications) | 1 (1) | 3 (4)
Procedural nausea (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Procedural pain (Injury, poisoning and procedural complications) | 41 (41) | 38 (38)
Dizziness (Nervous system disorders) | 6 (6) | 2 (2)
Headache (Nervous system disorders) | 3 (3) | 7 (7)
Insomnia (Psychiatric disorders) | 3 (3) | 1 (1)
Bladder spasm (Renal and urinary disorders) | 4 (4) | 4 (4)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In case a proposed publication contains reference to an invention owned by the sponsor or to which the sponsor otherwise has rights, the sponsor may request a reasonable suspension of the publication.